CLINICAL TRIAL: NCT04660123
Title: A Real World Study of Bismuth Colloidal Pectin Granules Quadruple Therapy for H. Pylori Eradication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Principal Investigator, Clinical Professor, Xijing Hospital of Digestive Diseases
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20202101-F-1
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Gastric Cancer; Helicobacter Pylori Infection; Bismuth
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quadruple therapy with colloidal bismuth pectin granules (Experimental): colloidal bismuth pectin granules 150 mg, Selection of 2 antibiotics and 1 proton pump inhibitor based on China's fifth national consensus report on the management of H. pylori infection.All medication is taken orally, twice a day.
  Interventions: Drug: Bismuth Colloidal Pectin Granules Quadruple Therapy for H. Pylori Eradication

INTERVENTIONS:
Drug: Bismuth Colloidal Pectin Granules Quadruple Therapy for H. Pylori Eradication — Standard dose of proton pump inhibitor, bismuth , and 2 antibiotics, 14 days course.
  Standard doses of proton pump inhibitors are esomeprazole 20mg, rabeprazole 10mg (or 20mg).
  Omeprazole 20mg, lansoprazole 30mg, pantoprazole 40mg, alprazole 5mg, any one of these.
  Bismuth is colloidal bismuth pellets, 150mg, 2 times/d.
  Antibiotic Program:
  Scheme 1 Amoxicillin 1000 mg, 2 times/d; Clarithromycin 500mg, 2 times per day Scheme 2 Amoxicillin 1000 mg, 2 times/d; Levofloxacin 5001 times/2 times Scheme 3 Amoxicillin 1000 mg, 2 times/d; Furazolidone 100mg, 2 times/d. Scheme 4 Amoxicillin 1000 mg, 2 times/d; Metronidazole 400mg, 3 times/d or 4 times/d Scheme 5 Amoxicillin 1000 mg, 2 times/d; Tetracycline 500mg, 3 times/d or 4 times/d Scheme 6 Tetracycline 500mg, 3 times/d or 4 times/d; Metronidazole 400mg, 3 times/d or 4 times/d Scheme 7 Tetracycline 500mg, 3 times/d or 4 times/d; Furazolidone 100mg, 2 times/d.

SUMMARY:
To observe the eradication rate of H. pylori infection, symptom improvement and the incidence of adverse effects in patients using a bismuth colloidal pectin granules quadruple therapy.

DETAILED DESCRIPTION:
The study will include three phases: screening, treatment and follow-up. Screening: Patients who have been screened to meet the criteria for naval platooning will be enrolled after signing an informed consent form.

Treatment: Subjects will receive 14 days of eradication treatment. With the exception of colloidal bismuth pectin granules, which will be limited, proton pump inhibitors (PPI) and 2 antibiotics will be selected on the basis of the physician's experience.

Follow-up: Includes two visits. approximately 14 days of treatment and 28 days after the end of treatment. Eradication of H. Pylori will be confirmed through urea breath test(UBT).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18~75,both gender.
2. Patients with upper gastrointestinal symptoms and with documented H.pylori infection.
3. Patients are willing to receive eradication treatment.
4. Women are eligible if they are not pregnant or nursing, and if they are of childbearing potential they are required to use medically acceptable contraception for the duration of the study and 30 days thereafter.

Exclusion Criteria:

1. Contraindications to study drugs.
2. Substantial organ impairment, severe or unstable cardiopulmonary or endocrine disease.
3. Constant use of anti-ulcer drugs ( including taking proton-pump.inhibitors(PPI) within 2 weeks before the [13C] urea breath test),antibiotics or bismuth complexes (more than 3 times /1 month before screening).
4. Patients were diagnosed with gastroduodenal ulcer and MALTlymphoma.
5. Pregnant or lactating women.
6. Underwent upper gastrointestinal Surgery.
7. Patients with Barrett esophageal or highly atypical hyperplasia, have symptom of dysphagia.
8. Evidence of bleeding or iron efficiency anemia.
9. A history of malignancy.
10. Drug or alcohol abuse history in the past 1 year.
11. Systemic use of corticosteroids, non steroidal anti-inflammatory drugs,anticoagulants, platelet aggregation inhibitors (except the use of aspirin for less than 100 mg/d).
12. Patients who has psychological problem or poor compliance.
13. Enrolled in other clinical trials in the past 3 months.
14. Refuse to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 959 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
helicobacter pylori eradication | 28 days after treatment
  The primary end point of this study is H.pylori eradication,established by negative [13C] urea breath test 28 days after the end of eradication.

SECONDARY OUTCOMES:
symptoms improvement rates | 14 days of treatment, and 28 days after treatment
  symptoms improvement rates Evaluation improvement rate of symptoms 2 weeks of treatment and 4 weeks after the end of treatment. Symptom improvement rate =#total score before treatment - total score after treatment#/total score before treatment x100%. Total score = frequency + severity.Frequency score is calculated by all the frequency of heartburn, reflux, abdominal pain, and flatulence, etc. Severity is accumulated by the degree of symptoms described above, which is divided to 4 degree as 0 presenting none, and 3 presenting most severe

OTHER OUTCOMES:
adverse events | 14 days of treatment, and 28 days after treatment
  Participants with Adverse Events as a Measure of Safety and Tolerability.The common side effects of the study include headache, dizziness, skin rash, other gastrointestinal disorders, pyrexia, cough and back pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China